CLINICAL TRIAL: NCT03893006
Title: On the Highway to Autonomous Driving: How is Automation Changing Humans: Investigations of Drivers' Behaviors, Representations and Neural Processes
Brief Title: Vehicle Automation Impact on Drivers
Acronym: AUTODRIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0141
Record Dates: First submitted 2019-03-08; First posted 2019-03-27 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Behaviors; Driving; Automation; Neuroimaging
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- UnAssisted (UA) (Experimental): This term refers to driving a vehicle manually without any vehicle automation technology. It will serve as a baseline concerning behaviors, representations and neural results associated with unassisted automobile driving.
  Interventions: Device: Level of vehicle automation
- Assisted (A) (Experimental): This term refers to driving with warning technology which upon activation sounds an a warning when the vehicle is too close to the edge of the road (off-road warning , Navarro, Mars, & Hoc, 2007; Suzuki & Jansson, 2003) or too close to the vehicle in front of it (anti-collision warning; Lee, McGehee, Brown, & Reyes, 2002).
  Interventions: Device: Level of vehicle automation
- Shared Control (SC) (Experimental): This term refers to shared tactical control between the driver and the automated assistive technology, both working simultaneously on the physical trajectory of the vehicle, laterally (Griffiths & Gillespie, 2005; Mulder, Abbink, & Boer, 2012) as well as longitudinal (Adell, Várhelyi, & Hjälmdahl, 2008).
  Interventions: Device: Level of vehicle automation
- Partly Autonomous (PA) (Experimental): This term refers to a situation where the lateral and longitudinal control of the driving are delegated to the automated assistive technology. It consists of a level of automatisation that today is possible to put into application and which often is referred to by the name "Highly Automated Driving" (Navarro, 2018). In this case, the driver is no longer the one who physically ensures the lateral and longitudinal control of the vehicle, but instead supervises the actions of the automated assistive technology.
  Interventions: Device: Level of vehicle automation
- Fully Autonomous (FA) (Experimental): This term refers to a completely automated driving experience. The on-board technologies take over all the driving tasks for any driving situation.
  Interventions: Device: Level of vehicle automation
- Any Automation (AA) (Experimental): This term refers to a situation where the drivers can choose the automation device of their choice among the five types presented above and can change it whenever they think it is good to do so.
  Interventions: Device: Level of vehicle automation

INTERVENTIONS:
Device: Level of vehicle automation — From no automation of the vehicle to full automation through warnings, shared control and partly automated automation levels.

SUMMARY:
In the context of ever-increasing automation in surface vehicles, automation impact on drivers will be investigated through three complementary research axes undertaken under simulated driving:

Axe 1 (Cognitive ergonomics), how automation is impacting driving behaviors and visual explorations? Axe 2 (Experimental psychology), how automation is impacting drivers' mental representations of their own driving abilities? Axe 3 (Neuroimaging), how automation is modifying the car driving neural network? And what are drivers' mental representations neural bases? The project tackle both applied and basic research issues using an original experimental neuro ergonomics approach. AUTODRIVE will bring original data on human-machine cooperation, mental representations, cognitive control and brain processes depending on the characteristics of the automation used over a significant period of time (six weeks) on a large sample (N=120) of experienced and inexperienced drivers.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 22 and 45 years old
* Having given an informed consent for the study
* Being registered with the French Social Security System
* No driving license for 60 participants
* Driving license for 4 years or more for 60 participants

Exclusion Criteria:

* No signature on the consent form
* Inability to read or write French.
* Neurologic or psychiatric illness, known or revealed during the inclusion visit
* Substance intake ( taking psychoactive medications or recreational drugs) on the day of the experiment
* Noise intolerance
* Need of vision glasses to drive
* Persons under curators or deprived of civil rights or deprived of their freedom
* Unable to fill a questionnaire (severe cognitive troubles)
* Subjects must not have metallic or electronic implants in the body : pacemakers or pacemaker wires, open heart surgery, artificial heart valve, brain aneurysm surgery, middle ear implant, hearing aid, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, or artificial limb or joint o foreign metallic objects in the body (bullets, BBs, pellets, shrapnel, or metalwork fragments) or current or past employment as machinists, welders or metal workers, tattoos near the head or neck regions, permanent makeup
* Claustrophobia

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-07-08 (Estimated); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
BOLD effect | Repetition Time (TR) :every 3 seconds, during the 3 fMRI sessions of respectively 1 hour, 0,75 hour and 0,75 hour. fMRI session 2 occurs 3 weeks after fMRI session 1 and 3 weeks before fMRI session 3.
  Functional magnetic resonance imaging measures brain activity by detecting changes associated with blood flow This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases. The primary form of fMRI uses the blood-oxygen-level dependent (BOLD) contrast in response to an experimental condition (Ogawa, Lee, Kay, & Tank, 1990), allowing researchers to track changes in oxygen consumption on the brain, and therefore brain activity. BOLD effect is computed by assessing the different relaxation times (T1 and T2) in the brain, as T1 and T2 are different in function of regional cerebral blood flows.
  The outcome will be a change between mean BOLD effect oven session 1 versus session 2 versus session 3.

SECONDARY OUTCOMES:
Behavioral changes | Two experimental sessions of an hour, one before and one after the six weeks of automated driving. Plus six driving sessions of 0,5 hour, one driving session the first day of each experimental week.
  Participants will be asked to drive through a variety of driving situations in a driving simulator simulated environment equipped with an eye-tracker. The measure collected will be drivers' behaviors on the steering wheel and pedals as well as their visual behaviors.
  The outcome will be a change in the number of actions on the steering wheel (a), pedals (b) and gaze dispersion (c) on the visual scene across the time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Navarro, MD, Principal Investigator — : Laboratoire d'Etude des Mécanismes Cognitifs (EMC) -Université Lumière Lyon 2
Locations (1):
- Laboratoire d'Etude des Mécanismes Cognitifs (EMC), Bron, France